CLINICAL TRIAL: NCT02650388
Title: Frailty and Cognitive Function Assessment of TAVI Patients (The Hungarian Frailty Score) - Observational, Prospective, Singe Center Study
Brief Title: Frailty and Cognitive Function Assessment of TAVI Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hungarian Institute of Cardiology (Other Government)
Collaborators: Semmelweis University (Other)
Responsible Party: Principal Investigator, ANDREKA PETER, Professor and Head of the department, Hungarian Institute of Cardiology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56174-1/2015/EKU(0470/15)
Record Dates: First submitted 2015-12-22; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Quality of Life; Aortic Valve Stenosis; Heart Valve Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases | interventions — Quality of Life; Walking Speed; Hand Strength; Activities of Daily Living; Serum Albumin; Mental Status and Dementia Tests; Wisconsin Card Sorting Test; Stroop Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post TAVI neurocognitive outcome (Other): TAVI with CoreValve will be done for all the patients and outcome will be assessed as Cognitive fuction, quality of life, Gait speed, Hand grip strength, Activities of daily living (ADL), Instrumental activities of daily living (IADL), Short- Form Mini Nutritional assessment (SF-MNA), Serum albumin level, Hemoglobin level, BMI, Montreal cognitive Assessment (MOCA), EQ-5D-3L-questionnaire, Ferreans and Powers Quality of life Index (QLI), MOCA, RBANS, Wisconsin test, Stroop test, Fluency test, Subjective "Eyeball test", Serial Transcranial Doppler (TCD) during TAVI. Finally, Hungarian frailty score will be deduced.
  Interventions: Behavioral: Cognitive fuction, quality of life

INTERVENTIONS:
Behavioral: Cognitive fuction, quality of life — To test the above score in patients undergoing TAVI
  Other Names: Gait speed; Hand grip strength; Activities of daily living (ADL); Instrumental activities of daily living (IADL); Short- Form Mini Nutritional Assessment (SF-MNA); Serum albumin level; Hemoglobin level; BMI; Montreal Cognitive Assessment (MOCA); EQ-5D-3L-questionnaire; Ferreans and Powers Quality of life Index (QLI); MOCA; RBANS; Wisconsin test; Stroop test; Fluency test; Subjective "Eyeball test"; Serial Transcranial Doppler (TCD) during TAVI

SUMMARY:
Aortic stenosis (AS) is the most common valve disease among the adult population, in the majority of the cases it only requires treatment in advanced age. Transcatheter aortic valve implantation (TAVI) has become available as an alternative treatment for very high risk or even inoperative patients who are suffering from symptomatic aortic stenosis. Until now it has been learnt that there are group of patients who are in a very bad condition and who are so frail that they do not benefit from TAVI. These patients have worse survival rate and more importantly poor quality of life in spite of a successful procedure. Cardiac surgery risk scores like Society of Thoracic surgery score (STS) and EUROSCORE are less accurate in aging high risk people. In elderly it is principal to make differentiation between utility and futility. On the other hand, beside frailty status the main barrier to TAVI is the risk of neurological impairment. Neurological injury and impairment in TAVI can occur as cerebrovascular event (CVE) and/or neurocognitive dysfunction. The two neurocognitive dysfunctions - post-operative delirium (POD) and post-operative cognitive dysfunction (POCD). Most cases remain undetected although clinically could be apparent or silent. The neurological injury can be observed and/or detected by neuroimaging techniques and cognitive trajectories. A well established and validated frailty score based on relatively simple and feasible tests could help in our everyday practice to evaluate the prognosis of elderly people undergoing TAVI and to determine those patients who really benefit from the procedure.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is the most common valve disease among the adult population, in the majority of the cases it only requires treatment in advanced age. Surgical aortic valve replacement (SAVR) is very often refused because of advanced age and poor general condition. These patients used to receive only medical treatment which is less favorable compared to SAVR. Nowadays transcatheter aortic valve implantation (TAVI) has become available as an alternative treatment for very high risk or even inoperable patients who are suffering from symptomatic aortic stenosis (1). Between 2012 and 2014 TAVI has been used extensively, accumulating over 100,000 procedures performed worldwide since 2002 (2). TAVI was originally developed for those patients who were considered too frail to undergo SAVR (3). Recently, we are able to perform TAVI in almost all patients with high procedure success rate and achieve good hemodynamic results. Despite these promising results, the one year outcome is not so evident. Until now it has been learnt that there are a group of patients who are in a very bad condition and who are so frail that they do not benefit from TAVI. These patients have worse survival rate and more importantly poor quality of life in spite of a successful procedure. Cardiac surgery risk scores like Society of Thoracic surgery score (STS) and EUROSCORE are less accurate in aging high risk people (4). Advanced age is often accompanied with frail general conditions and, the estimated morbidity and mortality values do not correlate well with the postoperative outcomes. In these risk scores very important relevant factors like frailty and disability are not taken into account. In elderly it is principal to make differentiation between utility and futility. Frailty is a clinical syndrome that reflects impaired physiologic reserve and increased vulnerability to stressors (5). However frailty as a geriatric concept has existed for a long time, its importance has recently gained high priority in the concept of older adults especially who undergo TAVI(1). By today frailty scores have increasing importance and are used more frequently by several investigators. Slow 5m gait speed has evidently proven unfavorable outcomes (6, 7), other frailty assessment tools like handgrip strength test, activities of daily living (ADL), instrumental activities of daily living (iADL), nutritional assessment, mini-mental status, etc. has been being investigated continuously.

On the other hand, beside frailty status the main barrier to TAVI is the risk of neurological impairment. The TAVI candidate patients have specific central nervous system (CNS) issues because of neurobiological changes of aging, e.g. decreased brain weight and volume, decreased neurotransmitter system function, decreased neuronal gene expression and Alzheimer type changes (8). Neurological injury and impairment in TAVI can occur as cerebrovascular event (CVE) and/or neurocognitive dysfunction. Both forms might be clinically apparent and detected, clinically apparent but undetected and clinically silent and undetected. The two neurocognitive dysfunctions - post-operative delirium (POD) and post-operative cognitive dysfunction (POCD) - most cases remain undetected although clinically could be apparent or silent (9). POD is defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). POCD is defined by Kappetein et al., as "deterioration of intellectual function presenting as impaired memory or concentration presenting with temporal association to surgery" (9, 10). The neurological injury can be observed and/or detected by neuroimaging techniques and cognitive trajectories. Some insult caused by TAVI might remain in the clinically silent area and might be observed only as slight neurocognitive dysfunction. Analization of the incidence and underlying etiology of the neurological events may lead to identification of recently non-recognized techniques or neuroprotective strategies, devices. The most elevated incidence of CVEs is within 24 hours of TAVI. This risk of further events might be high for up to two months (11). One fifth of health-related quality of life (HRQOL) is characterized by cognitive functions. Studies and reports on cognitive, psychiatric, and/or neurological events following TAVI have focused on major and well-marked complications, e.g., stroke, TIA, and post-operative delirium (12). Meantime TAVI is associated with a high incidence (73%-84%) of silent cerebral embolism as detected by diffusion-weighted MRI (13).

Chronological age does not always reflect biological age and there is a wide range between fit to frail (14). A well established and validated frailty score based on relatively simple and feasible tests could help in our everyday practice to evaluate the prognosis of elderly people undergoing TAVI and to determine those patients who really benefit from the procedure. Post-Operative Cognitive Dysfunction (POCD) in patients undergoing TAVI (and/or SAVR) was examined in only a few studies published during the last 10 years. Examinations and investigation of finer, long-term and possibly positive post-operative cognitive outcomes following TAVI (and SAVR) are significantly under-represented in the current medical literature (15).

Hypothesis:

There is a significant correlation between the Hungarian Frailty Score (HFS) and post procedure outcomes and quality of life preservation. HFS score would be a useful tool to estimate those who will benefit from TAVI. We also hypothesize that cognitive performance will be preserved, and will improve at the end of 12th month after TAVI due to better cerebral circulation.

Objectives and aims

1. Generate and validate a new risk score system called the Hungarian Frailty Score (HFS), which represents an objective tool for evaluation of the frailty syndrome in patients undergoing TAVI procedure.
2. To determine the changes and to prove that there is no cognitive decline in patients undergoing TAVI if so any (pre and post TAVI cognitive function will be assessed).

Primary aims:

To estimate the correlation between the HFS, and the in-hospital stay, 30 day and 1-year outcomes evaluated according to the VARC 2 Criteria. The benefit of this study is to conclude exact data about quality of life and provide a comprehensive investigation of pre- and post-TAVI cognitive outcomes. We plan to define that apart from the incidence of possible neurological signs and the radiological evidences of neurogical injury and POCD, there is no decline in long term cognitive functions and there is improvement in the long term quality of life (QoL).

Secondary aims:

Find correlation and differences between HFS, QoL, eyeball test, and cognitive outcomes. Additional impact is to assess whether POD and POCD are a part of same condition, spectrum, and what can we do to prevent them.

Expected results:

To generate a simple and useable risk score system adopted to the Hungarian population for evaluating patients who undergo TAVI and collect data about post TAVI QoL and cognitive functions, and to register changes in the pre and post procedure frailty score. Non-diagnosed preoperative cognitive impairments and CVEs of the patient will be detected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years,
* Severe, symptomatic aortic stenosis,
* High risk for cardiac surgery (STS and logistic Euroscore ),
* According multidisciplinary (heart) team decision TAVI is preferable,
* Willing to participate

Exclusion Criteria:

* Died before TAVI
* Not willing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
To correlate HFS with mortality at 30 days and 1-year | 1 year

SECONDARY OUTCOMES:
Find correlation and differences between HFS and QoL | 1 year
Find correlation and differences between HFS and eyeball testing | 1 year
Find correlation and differences between HFS and cognitive outcomes. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Andreka, MD, PhD., Principal Investigator — Hungarían Institute of Cardiology
Locations (1):
- Hungarian Institute of Cardiology, Budapest, Budapest, Hungary